CLINICAL TRIAL: NCT02319499
Title: Zinc, Iron and Vitamin A Supplementation for Infant Growth and Development, and the Contributing Role of Psychosocial Care
Brief Title: Zinc, Iron, Vitamin A and Psychosocial Care for Child Growth and Development
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Umi Fahmida, Dr, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ZIAP
Record Dates: First submitted 2014-12-07; First posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Development; Iron Deficiency; Zinc Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Zinc; Iron; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Zinc Alone (Experimental): Zinc Sulphate (10 mg Zn/day)
  Interventions: Dietary Supplement: Zinc Alone
- Iron and Zinc (Experimental): Ferrous Sulphate and Zinc Sulphate (10 mg/day of each zinc and iron)
  Interventions: Dietary Supplement: Iron and Zinc
- Iron, Zinc and Vitamin A (Experimental): Ferrous Sulphate, Zinc Sulphate and Vitamin A (10 mg/day of each zinc and iron, plus 1,000 IU vitamin A/day)
  Interventions: Dietary Supplement: Iron, Zinc and Vitamin A
- Placebo (Placebo Comparator): No minerals/vitamin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc Alone — Zn-alone group received 10 mg/day of elemental zinc (as zinc sulphate)
  Arms: Zinc Alone
Dietary Supplement: Iron and Zinc — Zn+Fe group received 10 mg/day of elemental zinc (as zinc sulphate) and 10 mg/day of elemental iron (as ferrous sulphate)
  Arms: Iron and Zinc
Dietary Supplement: Iron, Zinc and Vitamin A — Zn+Fe+vit.A group received 10 mg/day of elemental zinc (as zinc sulphate) and 10 mg/day of elemental iron (as ferrous sulphate), plus 1,000 IU/day of vitamin A
  Arms: Iron, Zinc and Vitamin A
Other: Placebo — Placebo group received no minerals/vitamin
  Arms: Placebo

SUMMARY:
Many Indonesian infants are already iron deficient before they reach the age of six months, which also determines the high prevalence of anemia among under-five children. Iron deficiency ultimately leads to anemia, and there is clear evidence that iron deficiency anemia during early childhood has a marked negative effect on child development and cognitive function (Lozoff et al.1991; Idjradinata & Pollitt, 1993). This negative impact on childhood development is one of the main reasons why iron deficiency during infancy should be prevented or treated.

Since diets low in iron is usually also low in zinc, zinc deficiency --which has negative consequence on growth-- is common in iron deficiency area. In Southeast Asia, the condition is exacerbated by the rich phytate content in the complementary foods which inhibits the absorption of iron as well as zinc (Gibson, 1994). Thus, combining both iron and zinc, hence, is expected to decrease both iron and zinc deficiencies and hence improve growth and development of the children.

Recently, there has been an emerging view which looks at the two-way relationship between nutrition, health, and psychosocial well-being. This concept is supported by studies on "positive deviance", a term used to refer to children who grow and develop well in impoverished environments where most children are victims of malnutrition and chronic illness (Zeitlin et al., 1990). The mechanism which helps to explain how psychosocial factors, such as the affect between mother and child, are associated with adequate growth and development: 'Psychological stress has a negative effect on the use of nutrients whereas psychological well-being stimulates the secretion of growth-promoting hormones. Pleasantly stimulating interactions can enhance the child's tendency to exercise its developing organ systems and hence to utilize nutrients for growth and development'.

Understanding how the psychosocial environment can promote or inhibit the benefit of supplementation intervention is necessary in order to have a better way of setting about providing supplements. In fact, many supplementation programs do not incorporate complementary program elements that would help to improve the health and psychosocial development of children at the same time that they improve nutritional status' (Myers, 1995). Looking from this perspective, not only will supplementation benefit the psychosocial development but also the psychosocial environment can promote the benefit of the supplementation on the nutritional status and developmental outcomes of infants.

The purpose of the study is to investigate whether multi-micronutrient supplementations (zinc+iron, zinc+iron+vit.A) have positive effect on infants' growth and developmental outcomes, and whether the effect is modified by psychosocial care.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 6 month old
* predominantly breast-fed children (assuming the infants were already introduced complementary feedings as early as 4 months)
* parental consent

Exclusion Criteria:

* apparent congenital abnormalities

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 1998-08; Primary Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Change in Length-for-Age Z-scores | Baseline and monthly thereafter until endline (6 month of intervention)
  Length-for-Age Z-score
Change in Weight-for-Length Z-scores | Baseline and monthly thereafter until endline (6 month of intervention)
  Weight-for-Length Z-score
Change in Weight-for-Age Z-scores | Baseline and monthly thereafter until endline (6 month of intervention)
  Weight-for-Age Z-scores
Changes in Mental Development Index | Baseline and Endline (6 month of intervention)
  MDI of Bayley Scale of Infant Development II
Changes in Psychomotor Development Index | Baseline and Endline (6 month of intervention)
  PDI of Bayley Scale of Infant Development II

SECONDARY OUTCOMES:
Changes in Hemoglobin | Baseline and Endline (6 month of intervention)
  measured for all subjects (200 per group)
Changes in serum zinc | Baseline and Endline (6 month of intervention)
  measured in sub-samples (65 subjects/group)
Changes in serum ferritin | Baseline and Endline (6 month of intervention)
  measured in sub-samples (65 subjects/group)
Changes in serum retinol | Baseline and Endline (6 month of intervention)
  measured in sub-samples (65 subjects/group)

CONTACTS AND LOCATIONS:
Overall Officials: Umi Fahmida, PhD, Principal Investigator — South East Asian Ministers of Education Organization, Regional Center for Food and Nutrition (SEAMEO-RECFON)
Locations (1):
- South East Asian Ministers of Education Organization, Regional Center for Food and Nutrition (SEAMEO-RECFON), Jakarta, Java, Indonesia

REFERENCES:
- [Background] Schultink W, Gross R. Iron deficiency alleviation in developing countries. Nutr Res Rev. 1996 Jan;9(1):281-93. doi: 10.1079/NRR19960015. No abstract available. PMID 19094274
- [Background] Colomer J, Colomer C, Gutierrez D, Jubert A, Nolasco A, Donat J, Fernandez-Delgado R, Donat F, Alvarez-Dardet C. Anaemia during pregnancy as a risk factor for infant iron deficiency: report from the Valencia Infant Anaemia Cohort (VIAC) study. Paediatr Perinat Epidemiol. 1990 Apr;4(2):196-204. doi: 10.1111/j.1365-3016.1990.tb00638.x. PMID 2362876
- [Background] Lozoff B, Brittenham GM, Wolf AW, McClish DK, Kuhnert PM, Jimenez E, Jimenez R, Mora LA, Gomez I, Krauskoph D. Iron deficiency anemia and iron therapy effects on infant developmental test performance. Pediatrics. 1987 Jun;79(6):981-95. PMID 2438638
- [Background] Idjradinata P, Pollitt E. Reversal of developmental delays in iron-deficient anaemic infants treated with iron. Lancet. 1993 Jan 2;341(8836):1-4. doi: 10.1016/0140-6736(93)92477-b. PMID 7678046
- [Background] Brown KH, Wuehler SE and Peerson JM (2001). The importance of zinc in human nutrition and estimation of the global prevalence of zinc deficiency. Food Nutr Bull 22 (2):113-25
- [Background] Gibson RS and Ferguson EL (1999). An Interactive 24-hour Recall for Assessing the Adequacy of Iron and Zinc Intakes in Developing Countries. ILSI Press, Washington DC
- [Background] Ronaghy HA, Reinhold JG, Mahloudji M, Ghavami P, Fox MR, Halsted JA. Zinc supplementation of malnourished schoolboys in Iran: increased growth and other effects. Am J Clin Nutr. 1974 Feb;27(2):112-21. doi: 10.1093/ajcn/27.2.112. No abstract available. PMID 4591425
- [Background] Walravens PA, Chakar A, Mokni R, Denise J, Lemonnier D. Zinc supplements in breastfed infants. Lancet. 1992 Sep 19;340(8821):683-5. doi: 10.1016/0140-6736(92)92229-9. PMID 1355797
- [Background] Umeta M, West CE, Haidar J, Deurenberg P, Hautvast JG. Zinc supplementation and stunted infants in Ethiopia: a randomised controlled trial. Lancet. 2000 Jun 10;355(9220):2021-6. doi: 10.1016/S0140-6736(00)02348-5. PMID 10885352
- [Background] Rosado JL, Lopez P, Munoz E, Martinez H, Allen LH. Zinc supplementation reduced morbidity, but neither zinc nor iron supplementation affected growth or body composition of Mexican preschoolers. Am J Clin Nutr. 1997 Jan;65(1):13-9. doi: 10.1093/ajcn/65.1.13. PMID 8988907
- [Background] Cavan KR, Gibson RS, Grazioso CF, Isalgue AM, Ruz M, Solomons NW. Growth and body composition of periurban Guatemalan children in relation to zinc status: a longitudinal zinc intervention trial. Am J Clin Nutr. 1993 Mar;57(3):344-52. doi: 10.1093/ajcn/57.3.344. PMID 8438768
- [Background] Bates CJ, Evans PH, Dardenne M, Prentice A, Lunn PG, Northrop-Clewes CA, Hoare S, Cole TJ, Horan SJ, Longman SC, et al. A trial of zinc supplementation in young rural Gambian children. Br J Nutr. 1993 Jan;69(1):243-55. doi: 10.1079/bjn19930026. PMID 8457531
- [Background] Engle P and Ricciuti HN (1995). Psychosocial aspects of care and nutrition. Food Nutr Bull 16(4):356-77
- [Background] Myers R (1995). The Twelve Who Survive: Strengthening Programmes of Early Childhood Development in the Thirld World. High/Scope Press, Michigan
- [Background] Bayley (1993). Bayley Scales of Infant Development: Manual, 2nd ed. Harcourt Brace & Co., San Antonio
- [Background] Caldwell BM and Bradley RH (1984). Home Observation for Measurement of the Environment. University of Arkansas, Little Rock - Arkansas